CLINICAL TRIAL: NCT00662337
Title: A Randomized, Two-Way Crossover Evaluation of the Bioequivalence Between Two Oral Formulations of Diphenhydramine: ULTRATAB Tablet Versus KAPSEALS Capsule
Brief Title: Bioequivalence Between Two Oral Formulations of Diphenhydramine Hydrochloride
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A2341003
Record Dates: First submitted 2008-03-20; First posted 2008-04-21 (Estimated); Last update posted 2011-09-08 (Estimated); Status verified 2011-09

CONDITIONS: Nasal Congestion
Keywords: Bioequivalence, diphenhydramine hydrochloride
MeSH Terms: conditions — Nasal Obstruction | interventions — Diphenhydramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Diphenydramine HCl
  Interventions: Drug: Diphenhydramine hydrochloride

INTERVENTIONS:
Drug: Diphenhydramine hydrochloride — After a ten-hour fast and a one-hour fluid restriction prior to each dosing period, subjects received supervised dosing of their first 25 mg treatment with approximately eight ounces of water. Following a seven-day washout, the comparison treatment was administered according to thye same procedure.
  Other Names: Benadryl Allergy; 25 mg KAPSEALS capsule; 25 mg ULTRATAB tablets

SUMMARY:
The purpose of this study is to determine if two formulations of diphenhydramine hydrochloride are bioequivalent.

DETAILED DESCRIPTION:
Subjects were required to observe a ten-hour fast and a one-hour fluid restriction prior to each dosing period.

Subjects were randomized into one of two active treatment groups, received supervised dosing of their treatment with approximately eight ounces of water, and were required to maintain fluid restriction for one hour after treatment. Following the one-hour post-dose fluid restriction, subjects could drink water, but consumer no other food or fluids for four hours post-dose.

Following a seven-day washout period, the comparison treatment was administered according to the same procedure as above.

ELIGIBILITY:
Inclusion Criteria:

* healthy male and/or female subjects between the ages of 18 and 55 years, inclusive
* approximately 18 to 30 kg/m2 BMI
* total body weight at least 55 kg (121 lbs)
* able to understand and sign the written Informed Consent Form
* willing to follow the protocol requirements and comply with protocol restrictions

Exclusion Criteria:

* pregnant or lactating women
* women of childbearing potential not using acceptable form of contraception 3 months prior to the first dose until completion of follow-up procedures
* history of allergy, sensitivity, and/or idiosyncratic reaction to Benadryl, diphenhydramine hydrochloride, or diphenhydramine citrate
* evidence of clinical, dietary or psychiatric deviation from normal that could increase the risk to the subject or research staff or interfere with the interpretation of study results
* use of licit or illicit drugs
* participated in any other trials within a specified number of days prior to the first dose of the trial treatment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2006-10; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence was assessed based on the pharmacokinetic variables, Cmax, AUC0-t and AUC0-infinity | At 15 minutes pre-dose (0 hour), and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 24, 36 and 48 hours post-dose

SECONDARY OUTCOMES:
The safety analysis included all subjects who took at least one dose of clinical trial test product and had any follow-up information. Subjects in the safety analysis set were summarized and listed, based on actual treatment received. | 15 minutes pre-dose (0 hour) through 28 days post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Israel, BS, Study Director — McNeil Consumer Healthcare Division of McNEIL-PPC, Inc.